CLINICAL TRIAL: NCT01703572
Title: A Phase 1 Dose Escalation Study of OMP-52M51 in Subjects With Lymphoid Malignancies
Brief Title: A Dose Escalation Study of OMP-52M51 in Subjects With Lymphoid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OncoMed Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mereo BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 52M51-001
Record Dates: First submitted 2012-09-27; First posted 2012-10-10 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Relapsed or Refractory Lymphoid Malignancies
Keywords: Phase 1; Dose escalation; relapsed or refractory; lymphoid malignancies
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OMP-52M51 (Experimental)
  Interventions: Drug: OMP-52M51

INTERVENTIONS:
Drug: OMP-52M51

SUMMARY:
This is an open-label Phase 1a dose escalation study of single-agent OMP-52M51 in subjects with relapsed or refractory lymphoid malignancies. Study includes a dose escalation phase and expansion phase. Subjects will be assessed for safety, immunogenicity, pharmacokinetics, biomarkers, and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Lymphoid malignancy that has relapsed or is refractory after two or more treatments that are FDA approved or are commonly used clinically.
2. Subjects must have progressive disease requiring therapy. Subjects who are candidates for observation only are not eligible.
3. Subjects are either not currently considered to be candidates or refuse potentially curative therapies including peripheral stem cell or bone marrow transplant
4. Subjects must have measurable disease as per disease specific criteria
5. Must have received their last chemotherapy, biologic, radiotherapy, or investigational therapy at least 4 weeks prior to enrollment; 12 weeks from their last radioimmunotherapy; 3 months if the last therapy was bone marrow/ peripheral stem cell transplant.
6. Age >18 years
7. ECOG performance status <2
8. Normal Ejection Fraction on ECHO scan
9. Subjects must have normal organ and marrow function as defined below:

   Absolute neutrophil count >1000/mL Platelets >75,000/mL For subjects with known marrow infiltration, ANC ≥500 and platelets ≥30,000 Total bilirubin <1.5 X institutional upper limit of normal (ULN) (<2X ULN for subjects with Gilbert's syndrome) AST (SGOT) and ALT (SGPT) <3 X institutional ULN (for subjects with hepatic involvement <5 X institutional ULN) PT/INR and aPTT within 1.5 X institutional ULN Creatinine <1.5 X institutional ULN OR Creatinine clearance >60 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal
10. Women of childbearing potential must have had a prior hysterectomy or have a negative serum pregnancy test and be using adequate contraception prior to study entry and must agree to use adequate contraception from study entry through at least 6 months after discontinuation of study drug. Men must also agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and from study entry through at least 6 months after discontinuation of study drug. Should a woman enrolled in the study or a female partner of a man enrolled in the study become pregnant or suspect she is pregnant while participating in this study or within 6 months after discontinuation of study, she should inform the Investigator immediately.
11. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

Subjects who meet any of the following criteria will not be eligible for participation in the study:

1. Currently receiving any therapeutic treatment for lymphoid malignancies including other investigational agents
2. Prior treatment with gamma secretase inhibitors or other Notch 1 inhibitors
3. Active CNS involvement, uncontrolled seizure disorder, or active neurologic disease
4. History of a Grade 4 allergic reaction attributed to humanized or human monoclonal antibody therapy
5. Significant intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
6. Pregnant women or nursing women
7. Ongoing malignancies or malignancies in remission <3 years other than the lymphoid malignancies included in this trial. Patients with history of known skin cancers including non-melanotic skin cancers within the past 3 years will not be included in this trial. The following prior malignancies are allowable irrespective of when they occurred: in situ carcinoma of the cervix, in situ ductal breast cancer, and low-grade local bladder cancer.
8. Subjects with known HIV infection
9. Known bleeding disorder or coagulopathy
10. Subjects receiving heparin, warfarin, or other similar anticoagulants, except for subjects on low molecular weight heparin for DVT/PE prophylaxis. Note: Subjects may be receiving low-dose aspirin and/or non-steroidal anti-inflammatory agents.
11. New York Heart Association Classification II, III, or IV
12. Subjects with a blood pressure of >140/90 mmHg that is not responsive to medical therapy. Subjects taking antihypertensive medications must be taking ≤2 medications to obtain this level of blood pressure control.
13. Subjects with EKG evidence of ischemia or ≥Grade 2 ventricular arrhythmia, subjects who have a history of acute myocardial infarction within 6 months, or subjects with unstable angina.
14. Subjects with known clinically significant gastrointestinal disease including, but not limited to, inflammatory bowel disease
15. Subjects with diarrhea at time of enrollment or have an ongoing requirement for anti diarrheal therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Safety profile of OMP-52M51 in subjects with relapsed or refractory lymphoid malignancies | Subjects will be assessed for DLTs from Days 0-29. Adverse events will be reported through 30 days after the last dose

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of OMP-52M51 in subjects with relapsed or refractory lymphoid malignancies | PK analyses at various time points following the 1st and 2nd doses, immediately pre and post-dose for all subsequent doses at treatment term, every 4 weeks after discontinuation of study drug or 12 weeks
  Apparent half life, AUC, clearance, volume of distribution
Immunogenicity of OMP-52M51 in subjects with relapsed or refractory lymphoid malignancies | At baseline, every 4 weeks, at treatment termination and every 4 weeks after the discontinuation of the study drug for 12 weeks.
Preliminary efficacy of OMP-52M51 in subjects with relapsed or refractory lymphoid malignancies | Evaluation for response will be assessed every 56 days and will be based on disease specific criteria.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of Colorado Hospital, Anschutz Cancer Pavilion, Aurora, Colorado
  - UF Health Davis Cancer Pavilion and Shands Med Plaza, Gainesville, Florida
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cornell University Division of Hematology and Medical Oncology, New York, New York
  - NYU Clinical Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Sara Cannon Research Institute, Nashville, Tennessee